CLINICAL TRIAL: NCT05363423
Title: Lateral Pedicled Nasoseptal Flaps for Endoscopic Draf III Procedure in Patients With Frontal Sinus Inverted Papilloma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TR-pedicled nasoseptal flaps
Record Dates: First submitted 2022-04-28; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Draf III Procedure; Naso-septal Flap; Inverted Papilloma
MeSH Terms: conditions — Papilloma, Inverted

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Procedure/Surgery: lateral pedicled nasoseptal flaps applied in Draf III procedure: The standard Draf III procedure was performed as described by Gross and Wormald using an "outside-in" technique. The cranial portion of the nasal septum was removed, and the frontal process of the maxilla and frontal beak were carefully abraded, resulting in the "frontal T". Distinct to the procedure of Gross and Wormald, the frontal T was then lowered to the first branch of the anterior ethmoidal artery instead of the first olfactory fibre. Tumors were totally resected under endoscope and lateral pedicled nasoseptal flaps were applied for covering the exposed bone around frontal neo-ostium. Type 1 flaps consisted of mucosa over the lateral nasal wall, and type 2 flaps consisted of the aforementioned mucosa and corresponding septal mucosa.
  Interventions: Procedure: Draf III procedure with lateral pedicled nasoseptal flaps applied
- Procedure/Surgery: no flaps applied in Draf III procedure: The standard Draf III procedure was performed as described by Gross and Wormald using an "outside-in" technique. The cranial portion of the nasal septum was removed, and the frontal process of the maxilla and frontal beak were carefully abraded, resulting in the "frontal T". Distinct to the procedure of Gross and Wormald, the frontal T was then lowered to the first branch of the anterior ethmoidal artery instead of the first olfactory fibre. Tumors were totally resected under endoscope and no flaps were applied.
  Interventions: Procedure: Draf III procedure without any flap applied

INTERVENTIONS:
Procedure: Draf III procedure with lateral pedicled nasoseptal flaps applied — The standard Draf III procedure was performed as described by Gross and Wormald using an "outside-in" technique. The cranial portion of the nasal septum was removed, and the frontal process of the maxilla and frontal beak were carefully abraded, resulting in the "frontal T". Distinct to the procedure of Gross and Wormald, the frontal T was then lowered to the first branch of the anterior ethmoidal artery instead of the first olfactory fibre. Type 1 flaps consisted of mucosa over the lateral nasal wall, and type 2 flaps consisted of the aforementioned mucosa and corresponding septal mucosa. After Draf III procedure, type 1 flaps were used to cover the bare bone of the ipsilateral frontal process and part of the ipsilateral anterior frontal table, which also constituted the bare bone area of the Draf II procedure. Type 2 flaps were used to cover for the bare bone of the ipsilateral frontal process and bilateral anterior or posterior frontal table.
  Groups: Procedure/Surgery: lateral pedicled nasoseptal flaps applied in Draf III procedure
Procedure: Draf III procedure without any flap applied — The standard Draf III procedure was performed as described by Gross and Wormald using an "outside-in" technique. The cranial portion of the nasal septum was removed, and the frontal process of the maxilla and frontal beak were carefully abraded, resulting in the "frontal T". Distinct to the procedure of Gross and Wormald, the frontal T was then lowered to the first branch of the anterior ethmoidal artery instead of the first olfactory fibre.
  Groups: Procedure/Surgery: no flaps applied in Draf III procedure

SUMMARY:
This is a retrospective case series study. The Draf III procedure exposes excessive bare bone, resulting in frontal ostium restenosis and surgical failure. For tumors originating from frontal sinus, especially inverted papillomas, abrading of bone around frontal ostium often exacerbate the restenosis. This study aims to retrospectly recruit patients with frontal sinus inverted papillomas who received Draf III procedure in our center during 2015-2021 and investigated the efficacy of a novel pedicled nasoseptal flap for endoscopic frontal sinus procedures. Each subject received a CT and magnetic resonance imaging (MRI) scans before operation. The subjects were followed up postoperative for at least 12 months to check the epithelization status and whether the neo-ostium were patent.

DETAILED DESCRIPTION:
The standard Draf III procedure was performed as described by Gross and Wormald using an "outside-in" technique. The cranial portion of the nasal septum was removed, and the frontal process of the maxilla and frontal beak were carefully abraded, resulting in the "frontal T". Distinct to the procedure of Gross and Wormald, the frontal T was then lowered to the first branch of the anterior ethmoidal artery instead of the first olfactory fibre.

Tumors were totally resected under endoscope and lateral pedicled nasoseptal flaps were applied for covering the exposed bone around frontal neo-ostium. The pedicled nasoseptal flaps were applied in the experimental group and no flap was applied in the control group.

The pedicle of the flap was designed to be on the frontal process of the lateral nasal wall. The lateral anterior incision was approximately 1 cm anterior to the maxillary line, with the medial anterior limit in parallel on the septum. The lateral posterior limit was the maxillary line and medial posterior limit parallel to the anterior limit where the first branch of the anterior ethmoidal artery arises on ethmoidal roof. The lower limit of the septal part was at the level of the lower border of the middle turbinate. The flap was carefully elevated from the cartilage and bone, particularly the supra-axillary and olfactory fossa part. The flap was then persevered posteriorly in the nasal floor or maxillary sinus for subsequent use. The contralateral flap was harvested and preserved in a similar manner. Type 1 flaps consisted of mucosa over the lateral nasal wall, and type 2 flaps consisted of the aforementioned mucosa and corresponding septal mucosa.

All patients were followed up for at least 12 months, and the nasal cavity was assessed and cleaned regularly under endoscopy. The neo-ostium section area was compared to that at the end of surgery. Epithelization was identified if the neo-ostium were smooth without edema, discharging or crusting after surgery under endoscope. The time required for epithelialization of each patient was also recorded. Restenosis was defined as >50% reduction in the section area at 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with bilateral frontal inverted papilloma who received a endoscopic endonasal Draf III surgery.
2. Ages range from 18-85 years old.
3. Preoperative CT and MRI scanning show favourable frontal sinus pneumatization.
4. Patients who are willing to following up regularly with good compliance.

Exclusion Criteria:

1. Patients who had undergone prior partial septectomy or septal perforation.
2. Patients who can't finish a regular 1-year follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with bilateral frontal inverted papilloma who received a endoscopic endonasal Draf III surgery between 2015 to 2021 in our center.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-10 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Time needed for epithelization | within 12 months postoperatively
  Epithelization was defined if the neo-ostium and the fused frontal sinus were smooth without edema, discharging or crusting after surgery under endoscope. Time needed for each subject was recorded.
Whether or not the frontal neo-ostium was restenosed | 12 months postoperatively
  Patients were checked under endoscope, and restenosis of neo-ostium was defined as a reduction of more than 50% in the section area compared to that at the end of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Study Chair — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
We haven't decided yet about the IPD sharing.

REFERENCES:
- [Background] Draf W. Endonasal micro-endoscopic frontal sinus surgery: The Fulda concept. Oper Tech Otolaryngol Head Neck Surg 1991; 2(4): 234-240.
- [Background] Lee JT, Kennedy DW, Palmer JN, Feldman M, Chiu AG. The incidence of concurrent osteitis in patients with chronic rhinosinusitis: a clinicopathological study. Am J Rhinol. 2006 May-Jun;20(3):278-82. doi: 10.2500/ajr.2006.20.2857. PMID 16871929
- [Background] Tran KN, Beule AG, Singal D, Wormald PJ. Frontal ostium restenosis after the endoscopic modified Lothrop procedure. Laryngoscope. 2007 Aug;117(8):1457-62. doi: 10.1097/MLG.0b013e31806865be. PMID 17585278
- [Background] Wormald PJ. Salvage frontal sinus surgery: the endoscopic modified Lothrop procedure. Laryngoscope. 2003 Feb;113(2):276-83. doi: 10.1097/00005537-200302000-00015. PMID 12567082
- [Background] Carney AS. Draf III frontal sinus surgery: "How I do it". Am J Rhinol Allergy. 2017 Sep 1;31(5):338-340. doi: 10.2500/ajra.2017.31.4458. PMID 28859713
- [Background] Abuzeid WM, Vakil M, Lin J, Fastenberg J, Akbar NA, Fried MP, Fang CH. Endoscopic modified Lothrop procedure after failure of primary endoscopic sinus surgery: a meta-analysis. Int Forum Allergy Rhinol. 2018 May;8(5):605-613. doi: 10.1002/alr.22055. Epub 2017 Dec 6. PMID 29210504
- [Background] DeConde AS, Smith TL. Outcomes After Frontal Sinus Surgery: An Evidence-Based Review. Otolaryngol Clin North Am. 2016 Aug;49(4):1019-33. doi: 10.1016/j.otc.2016.03.024. PMID 27450618
- [Background] Conger BT Jr, Riley K, Woodworth BA. The Draf III mucosal grafting technique: a prospective study. Otolaryngol Head Neck Surg. 2012 Apr;146(4):664-8. doi: 10.1177/0194599811432423. Epub 2012 Jan 6. PMID 22228601
- [Background] Deconde AS, Vorasubin N, Thompson CF, Suh JD. Rotation flaps after Draf procedures: a cadaver study. Otolaryngol Head Neck Surg 2012; 147(2): P255-P255.